CLINICAL TRIAL: NCT01125150
Title: Spectroscopic and Colorimetric Analysis of Acanthosis Nigricans in Patients With Hyperinsulinemia
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Dermatologist, Henry Ford Health System
Other Study IDs: IRB5339
Record Dates: First submitted 2010-05-12; First posted 2010-05-18 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2010-05

CONDITIONS: Acanthosis Nigricans; Hyperinsulinemia; Spectroscopic Analysis
Keywords: diffuse reflectance spectroscopy
MeSH Terms: conditions — Acanthosis Nigricans; Hyperinsulinism | interventions — Metformin; Diet Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Metformin — Dosage to be determined by Endocrinologist
Behavioral: Dietary Modification — To be determined by Endocrinologist

SUMMARY:
Acanthosis Nigricans is skin disease that associated with hyperinsulinemia. Clinical is velvety hyperpigmented plaques on neck, axilla, groin. If hyperinsulinemia is improved by treated with oral metformin and/ or diet control, acanthosis nigricans would be improved as well. Hyperpigmented plaques will be changed. We assess objective measurement by using spectroscopic and colorimetric analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have an elevated fasting insulin level, suggesting they are in an insulin resistant state.
2. Subjects must carry a diagnosis of acanthosis nigricans, which will be verified by a Dermatologist before entry into the study. If necessary, a small 4mm punch biopsy may be taken to document dermatopathology consistent with acanthosis nigricans.
3. Subjects must be willing and able to undergo treatment with Metformin, including initial referral and follow up.
4. Agree to abide by the investigator's guidelines
5. Be able to understand the requirements of the study, the risks involved and are able to sign the informed consent form
6. Agree to follow and undergo all study-related procedures

Exclusion Criteria:

1. Subjects with Type 1 Diabetes are excluded because of their naturally insulin-deficient, rather than hyper-insulinemic, states.
2. Women who are lactating, pregnant, or planning to become pregnant.
3. Any reason the investigator feels the patient should not participate in the study.

   -

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with both hyperinsulinemia and acanthosis nigricans.
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2009-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iltefat Hamzavi, M.D., Principal Investigator — Department of Dermatology, Henry Ford Hospital
Locations (1):
- Department of Dermatology, NEW CENTER ONE, Detroit, Michigan, United States